CLINICAL TRIAL: NCT05938816
Title: Feasibility and Acceptability of Stress Induction, Physiological Data Collection, and Mindfulness-Based Stress Reduction Among Combat Veterans With PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI change of career
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon Clinical and Translational Research Institute (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Joshua Kaplan, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00025508; KL2TR002370 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-07-10 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Ptsd
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness-Based Stress Reduction; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Health and Wellness Education (Placebo Comparator)
  Interventions: Behavioral: Health and Wellness Education (HWE)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — MBSR consists of weekly two-hour sessions for eight weeks, and a 7.5 hour retreat between weeks 6 and 7. The MBSR intervention will be facilitated by an experienced and certified MBSR teacher. MBSR curriculum strongly encourages completion of home practice assignments (~30 minutes daily) to help integration of concepts into daily life. Participants will receive audio CDs and a DVD to help guide home practice.
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Health and Wellness Education (HWE) — HWE is a didactic-based group intervention designed as an active comparator for randomized-controlled trials of MBSR. HWE provides instruction to participants regarding improving their emotional and physical health. In contrast to MBSR, there are no attempts to train participants' breathing, movement, or meditation habits or practices. HWE is administered in 8 weekly 2.5-hour classes with home practice to be completed between sessions (matched to MBSR for amount and effort). HWE also features one extended 7.5-hour retreat, similar to MBSR.84 Dr. Autumn Gallegos (consultant) has conducted trials of MBSR among veterans with PTSD using a HWE control group, and will provide mentorship to the PI in administering the HWE intervention. Dr. Kaplan and a trained RA will facilitate HWE.
  Arms: Health and Wellness Education

SUMMARY:
Investigators will recruit up to 20 veterans with PTSD. Participants will be randomized into two conditions: MBSR and Health and Wellness Education (HWE; control group). Participants will be randomized at a 1:1 ratio. Purpose of the study is to learn how mindfulness meditation may be helpful in treating PTSD. Participants will undergo 2 screening sessions, 8 weekly sessions of intervention (MBSR or HWE), 3 laboratory visits that will include completing survey questionnaires, stress test and recording of heart rate, blood pressure and breathing rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-85yo)
* Military veteran
* Experiencing PTSD symptoms
* Reading and speaking in English
* Be able to travel to OHSU for three two-hour lab visits, 8 weekly intervention sessions and one long extended session, and a two- hour focus group

Exclusion Criteria:

* Pregnancy
* Severe untreated depression, cognitive impairment, or active suicidality*
* Life-threatening or severely disabling medical conditions
* Excessive use of alcohol, nicotine, or cannabis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Kaplan, PhD, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants screened eligible and were consented. However no participants were assigned to arms, and no participants began study interventions or received treatment due to closure of study resulting from PI career change.
Period: Overall Study
Arm/Group | Mindfulness-Based Stress Reduction | Health and Wellness Education
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data not collected due to study being concluded prematurely due to PI change of career.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Stress Reduction | Health and Wellness Education | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Interview Targeting Feasibility of MBSR
Description: Qualitative data generated via focus group interviews. Questions will include common barriers to completing the intervention and strategies utilized by participants to maximize adherence.
Time Frame: 2 weeks post conclusion of intervention
Population: Data were not collected due to prematurely study closure due to PI change of career.
Arm/Group | Mindfulness-Based Stress Reduction | Health and Wellness Education
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Qualitative Interview Targeting Acceptability of MBSR
Description: Qualitative data generated via focus group interviews. Questions will include ratings of the relevance of the content presented to participants' lives, as well as assessment of the method of presentation.
Time Frame: 2 weeks post conclusion of intervention. Data were not collected due to prematurely study closure due to PI change of career.
Reporting Status: Not Posted

3. Secondary Outcome: Psychological Resilience 1
Description: Measured by self-report measure: Brief Resilience Scale (BRS). Scale ranges from 1-5 and higher scores indicate higher psychological resilience.
Time Frame: Pre (week 0), mid (week 4), and post intervention (week 10). Data were not collected due to prematurely study closure due to PI change of career.
Reporting Status: Not Posted

4. Secondary Outcome: Blood Pressure Reactivity
Description: Reactivity of physiological parameters (e.g., systolic and diastolic blood pressure) to a cognitive stress task.
Time Frame: Pre (week 0), mid (week 4), and post intervention (week 10).
Reporting Status: Not Posted

5. Secondary Outcome: PTSD Symptoms 1
Description: Measured by a self-report questionnaire: the PTSD Symptom Checklist (PCL). Scores range from 0-4 and higher scores indicate more severe PTSD symptoms.
Time Frame: Pre (week 0), mid (week 4), and post intervention (week 10).
Reporting Status: Not Posted

6. Secondary Outcome: Psychological Resilience 2
Description: Measured by self-report measure: Connor-Davidson Resilience Scale (CD-RISC). Scores range from 0-4 and higher scores indicate higher psychological resilience.
Time Frame: Pre (week 0), mid (week 4), and post intervention (week 10).
Reporting Status: Not Posted

7. Secondary Outcome: PTSD Symptoms
Description: Measured a clinician-administered semi-structured interview: the Clinician-Administered PTSD Scale (CAPS-5). Symptoms are rated for severity (0-absent; 1-mild/subthreshold; 2-moderate/threshold; 3-severe/markedly elevated; 4-extreme/incapacitating) and the presence of distress (minimal; clearly present; pronounced; extreme). Symptom clusters are also rated for the likelihood that they are related to the index trauma (definite; probable; unlikely).
Time Frame: Pre (week 0), mid (week 4), and post intervention (week 10).
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The study used the clinicaltrials.gov definition of adverse event and/or serious adverse event.
  Study was closed prior to randomization; therefore, no adverse events were collected or reported.
Arm/Group | Mindfulness-Based Stress Reduction | Health and Wellness Education
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT05938816/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT05938816/ICF_001.pdf